CLINICAL TRIAL: NCT02793414
Title: Diagnostic Utility of Volatile Organic Compounds in Human Breath for Acute Clinical Malaria in Ethiopia
Status: Withdrawn | Type: Observational
Sponsor: Menzies School of Health Research (Other)
Responsible Party: Sponsor
Other Study IDs: VOCE
Record Dates: First submitted 2016-05-26; First posted 2016-06-08 (Estimated); Last update posted 2020-10-06 (Actual); Status verified 2020-10

CONDITIONS: Malaria
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Malaria patients
- Febrile controls

SUMMARY:
This is a diagnostic efficacy study to evaluate a set of biomarkers in human breath indicative of an acute malaria infection. The investigators plan to enroll 75 malaria patients and 175 febrile non-malaria patients in Ethiopia.

Upon enrollment, blood for malaria RDT, microscopy and PCR will be collected as well as a breath sample to assess the presence of biomarkers at a reference center. Malaria patients identified by microscopy are revisited at day 2 and 7 to collect a further samples. G6PD testing will be performed concurrently to identify prevalent G6PD variants.

ELIGIBILITY:
Malaria cohort

* Age ≥5 years of age
* Malaria microscopy and / or Malaria RDT confirmed malaria infection
* Fever (axillary temperature ≥37.5⁰C) or history of fever in preceding 48 hours
* Written informed consent Febrile controls
* Age ≥5 years of age
* Fever (axillary temperature ≥37.5⁰C) or history of fever in preceding 48 hours
* Absence of a malaria episode confirmed by malaria microscopy
* Written informed consent

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Any participant above the age of 5 years fulfilling the inclusion criteria and attending the study hospital is eligible to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2016-09; Primary Completion 2017-04 (Estimated); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Performance of the VOC breathalyser | 7 days
  Sensitivity and specificity of the VOC breathalyser compared to microscopy, rapid diagnostic tests (RDTs) and PCR for the diagnosis of clinical malaria.

SECONDARY OUTCOMES:
Correlation of malaria parasite density with VOC concentrations | 7 days
  The correlation of malaria parasite density with VOC concentrations in patients with clinical and subpatent malaria and the recovery profile of VOC following acute malaria.
G6PD variants | 1 day
  G6PD variants within the local population
G6PD activity in U/gHb | 1 day
  The distribution of G6PD enzyme activity in the local population measured in U/gHb.
Performance characteristics of qualitative and quantitative G6PD test formats. | 1 day
  Sensitivity and specificity of other G6PD diagnostic assays compared to the gold standard spectrophotometry